CLINICAL TRIAL: NCT06298617
Title: Systemic Inflammatory Indices as a Non-invasive Grading Modality for Endometriosis: A Comparative Study Versus Exploratory Laparoscopy
Brief Title: Systemic Inflammatory Indices as a Non-invasive Grading Modality for Endometriosis
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Sabra, Lecturer of Obstetrics & Gynecology Department, Faculty of Medicine., Benha University
Other Study IDs: RC 27.1.2024
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy; Blood Cell Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Procedure: Diagnostic laparoscopy; Diagnostic Test: Full Blood Count (FBC)

INTERVENTIONS:
Procedure: Diagnostic laparoscopy — All women will undergo exploratory laparoscopy under general anesthesia
Diagnostic Test: Full Blood Count (FBC) — Blood samples withdrawn from patients on EDITA tubes and gone through full blood count and differential leucocytic count

SUMMARY:
Endometriosis (EMs) is one of the commonest chronic inflammatory disorder affecting women and is characterized by the presence and growth of endometrial-like glandular epithelial and stromal cells outside the uterus leading to multiple clinical symptoms affecting patients quality of life and fertility with high recurrence rate . The systemic immune inflammatory index (SII) and systemic inflammatory response index (SIRI) are documented as prognostic serum biomarker in many kinds of cancer and for the need and outcomes of adjuvant therapies for various cancers .

ELIGIBILITY:
Inclusion Criteria:

* Women with clinical manifestations suggestive of having EM;
* Women who was professionally diagnosed;
* Women who was diagnosed by radiologic workup;
* Women were free of exclusion criteria.

Exclusion Criteria:

* Women with EM and were maintained on treatment or underwent operative interference during the last three months;
* Patients had autoimmune diseases, maintained on immunosuppressive therapy for any indication;
* Women with cancer elsewhere in the body or receiving adjuvant therapies for cancer;
* Patients receiving therapies for viral disorders especially COVID;
* Patients refusing to undergo the exploratory laparoscopy.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women attending the outpatient of Gynecology department with clinical picture suggestive of having EM or had previously diagnosed depending on radiologic workup were evaluated for the enrolment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Indices' ability to predict EM stage | 8 months
  Number of patients was diagnosed with EM and got staged right through a calculated indices to the patients who went for exploratory laparoscopy which improve the chances of calculated indices facing the laparoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Al Qalyobia, Egypt